CLINICAL TRIAL: NCT04927559
Title: Assessing Health Literacy and Interpreter Use in Radiation Oncology at LAC+USC Medical Center
Brief Title: Health Literacy in Understanding Radiation Therapy Information in Patients Undergoing Definitive Radiation Therapy
Status: Terminated | Type: Observational
Why Stopped: Low accrual
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 0S-20-6; NCI-2020-06668 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 0S-20-6 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2021-05-25; First posted 2021-06-16 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage IA Breast Cancer AJCC v8; Anatomic Stage IB Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage IIA Breast Cancer AJCC v8; Anatomic Stage IIB Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Prognostic Stage I Breast Cancer AJCC v8; Prognostic Stage IA Breast Cancer AJCC v8; Prognostic Stage IB Breast Cancer AJCC v8; Prognostic Stage II Breast Cancer AJCC v8; Prognostic Stage IIA Breast Cancer AJCC v8; Prognostic Stage IIB Breast Cancer AJCC v8; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8; Stage I Prostate Cancer AJCC v8; Stage II Prostate Cancer AJCC v8; Stage IIA Prostate Cancer AJCC v8; Stage IIB Prostate Cancer AJCC v8; Stage IIC Prostate Cancer AJCC v8; Stage III Prostate Cancer AJCC v8; Stage IIIA Prostate Cancer AJCC v8; Stage IIIB Prostate Cancer AJCC v8; Stage IIIC Prostate Cancer AJCC v8; Stage IVA Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational (survey): Patients complete a survey over 5-10 minutes about their understanding of radiation therapy.
  Interventions: Other: Survey Administration

INTERVENTIONS:
Other: Survey Administration — Complete survey

SUMMARY:
This study assesses the health literacy and understanding of radiation therapy information during consultation in patients with prostate or breast cancer undergoing definitive radiation therapy. Health literacy is defined as "the capacity to obtain, process, and understand health information and services to enable sound health decisions." Information gained from this study, may help researchers develop appropriate modalities to enhance comprehension of radiation therapy, and therefore allow for improved patient decision making with medical treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess patient health literacy and understanding of critical radiation information during consultation in Spanish and English speaking patient in the department of radiation oncology at Los Angeles County (LAC) + University of Southern California (USC) utilizing a patient survey administered after consultation.

SECONDARY OBJECTIVE:

I. Correlate findings of radiation comprehension and satisfaction with validated measures of health literacy, acculturation, and socioeconomic status of patients.

TERTIARY OBJECTIVE:

I. To assess patient satisfaction of interpreter service in Spanish-speaking patients among breast and prostate cancer patients receiving definitive radiation.

OUTLINE:

Patients complete a survey over 5-10 minutes about their understanding of radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* All participants in this study will have cT1-4N0-1M0 prostate cancer or cT1-4N1-3M0 breast cancer, as clinically staged by the attending radiation oncologist following the American Joint Committee on Cancer (AJCC) 8th edition
* Non-metastatic breast or prostate cancer
* Radiation consultation for definitive treatment
* English or Spanish-speaking

Exclusion Criteria:

* Any person with major cognitive deficit or psychiatric impairment
* Any person, who with assistance by a family member or caregiver, is unable to complete a written survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: English and Spanish-speaking patients receiving care through LAC + USC radiation oncology who are being seen in consultation for definitive radiation for breast or prostate cancer.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2024-04-23 (Actual); Study Completion 2024-04-23 (Actual)

PRIMARY OUTCOMES:
Understanding of radiation therapy information | Up to 1 week
  Patients will be given an internally developed questionnaire of 11 questions intended to ascertain understanding of basic radiotherapy information that is needed to make an informed decision. The questions with one answer will be given a +1 for correct and -1 for incorrect. The questions with multiple answers (toxicity) will be given a +1 for a correctly chosen side effect, and a -1 for an incorrect response. The total will be the patient's summary score.

SECONDARY OUTCOMES:
Radiation comprehension and satisfaction | Up to 1 week
  Findings will be correlated with validated measures of health literacy, acculturation, and socioeconomic status of patients. Will assess variables associated with post-consult knowledge, with independent variables (IVs) comprising of ethnicity, cultural factors (nativity, acculturation), level of health literacy, sex, and socioeconomic status in linear regression models. Bivariate analyses will initially be conducted between IVs and the outcome; variables that are significant at p < 0.10 will be included in the multivariable model. Interaction terms will also be examined to test for differences by Hispanic/non-Hispanic ethnicity (the outcome regressed on Hispanic*IVs). The alpha level for the multivariable model will be p < 0.05.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Miller, MD, Principal Investigator — University of Southern California
Locations (1):
- Los Angeles County-USC Medical Center, Los Angeles, California, United States